CLINICAL TRIAL: NCT04334629
Title: Lipid Ibuprofen Versus Standard of Care for Acute Hypoxemic Respiratory Failure Due to COVID-19: a Multicentre, Randomised, Controlled Trial
Brief Title: LIBERATE Trial in COVID-19
Acronym: LIBERATE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn.
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 282009
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus; Respiratory Distress Syndrome; SARS-CoV Infection
MeSH Terms: conditions — Coronavirus Infections; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention)
- Standard of care plus lipid ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Lipid ibuprofen 200 mg
  Other Names: Flarin
  Arms: Standard of care plus lipid ibuprofen

SUMMARY:
The study aims to evaluate the reduction in severity and progression of lung injury with three doses of lipid ibuprofen in patients with SARS-CoV-2 infections.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years and above;
2. Hospitalised;
3. Confirmed or suspected SARS-CoV-2 infection;
4. National Early Warning Score (NEWS2) greater than or equal to 3 in a single parameter or NEWS2 > 5 overall;
5. Acute hypoxemic respiratory failure: PaO2/FiO2 ratio less than or equal to 300 OR SpO2/FiO2 ratio < 315 (Kigali Modification)
6. Provision of written informed consent by the patient OR by the patient's Legal Representative OR professional consultee.

Exclusion Criteria:

1. Any of the following contraindications to ibuprofen:

   * A known hypersensitivity to ibuprofen or any other constituent of the medicinal product;
   * Patients who have previously shown hypersensitivity reactions (e.g. asthma, rhinitis, angioedema or urticaria) in response to aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs);
   * Patients with a history of, or existing gastrointestinal ulceration/perforation or bleeding, including that associated with NSAIDs;
   * Patients with severe hepatic failure;
   * Patients with acute renal failure;
   * Patients with severe heart failure.
2. Participation in any other investigational drug products less than 30 days prior to study enrolment;
3. Glasgow Coma Score < 12;
4. Patients who cannot swallow oral capsules;
5. Pregnant or lactating women;
6. Any medical history that might, in the opinion of the attending clinician, put the patient at significant risk if he/she were to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Disease progression | 14 days
  Worsening respiratory failure; defined using severity of hypoxaemia using [PaO2/FiO2 ratio OR SpO2/FiO2 ratio]
Time to mechanical ventilation | 14 days
  Time to mechanical ventilation (or need of)

SECONDARY OUTCOMES:
Overall survival | 28 days
Reduction in proportion of patients who require ventilation | 28 days
Reduction in length of Critical Care stay | 28 days
Reduction in length of Hospital stay | 28 days
Modulation of serum pro- and anti-inflammatory cytokines | 28 days
Reduction in duration of ventilation | 28 days
Increase in ventilator-free days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Beale, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided